CLINICAL TRIAL: NCT00948012
Title: Exercise-induced Pulmonary Hypertension in Patients With Sickle-cell Anemia: an Echocardiographic Study.
Brief Title: Exercise-induced Pulmonary Hypertension in Patients With Sickle-cell Anemia
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Newton Nunes de Lima Filho, Federal University of São Paulo
Other Study IDs: HPSC01
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Sickle Cell Anemia; Pulmonary Hypertension
Keywords: Sickle Cell Anemia; Pulmonary Hypertension; Exercise echocardiography; Echocardiography
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients without pulmonary hypertension: Patients with sickle cell with normal response of pulmonary artery pressure to exercise
- Exercise-induced pulmonary hypertension: Patients with sickle-cell anemia with exercise-induced pulmonary hypertension.

SUMMARY:
Pulmonary hypertension (PH) at rest is a risk factor for death in patients with sickle-cell anemia (SCA). Exercise echocardiography (EE) can detect latent PH. We sought to investigate the occurrence of exercise-induced PH in patients with SCA and normal pulmonary pressure (PP) at rest, and its relationship with clinical and echocardiographic variables.Forty-four patients with SCA and normal PP at rest were studied and divided into two groups: exhibiting normal PP after treadmill EE (TRV≤2.7m/s) (G1), and exhibiting exercise-induced PH (TRV>2.7m/s) (G2). TRV cutoff points at rest and during exercise were based on data from healthy control subjects, matched for age, sex, and body surface area. Data obtained from EE were correlated with clinical, echocardiographic and ergometric variables.Exercise-induced PH occurred in 57% of the sample (G2), significantly higher than those of G1. Exercise-induced PH was related to higher levels of creatinine (p<0.05), increased left atrial volume (p<0.05) and right ventricular diastolic area (p<0.05), larger E/Em waves ratio derived from spectral and tissue Doppler (p<0.05), and higher TRV at rest (p<0.005).We concluded that patients with SCA and normal PP at rest may exhibit exercise-induced PH, which was related to renal function, increased cardiac chambers, abnormal indices of diastolic function and baseline TRV levels.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) at rest is a risk factor for death in patients with sickle-cell anemia (SCA). Exercise echocardiography (EE) can detect latent PH. We sought to investigate the occurrence of exercise-induced PH in patients with SCA and normal pulmonary pressure (PP) at rest, and its relationship with clinical and echocardiographic variables.Forty-four patients (22 men, mean age 25 y.o.) with SCA and normal PP at rest (tricuspid regurgitant jet flow velocity [TRV] <2.5 m/s) were studied and divided into two groups: exhibiting normal PP after treadmill EE (TRV≤2.7m/s) (G1), and exhibiting exercise-induced PH (TRV>2.7m/s) (G2). TRV cutoff points at rest and during exercise were based on data from healthy control subjects, matched for age, sex, and body surface area. Data obtained from EE were correlated with clinical, echocardiographic and ergometric variables.Exercise-induced PH occurred in 57% of the sample (G2), with mean TRV level of 3.4±0.4 m/s (range 2.8 - 4.5m/s), significantly higher than those of G1 (2.5±0.3 m/s, p<0.001). Exercise-induced PH was related to higher levels of creatinine (p<0.05), increased left atrial volume (p<0.05) and right ventricular diastolic area (p<0.05), larger E/Em waves ratio derived from spectral and tissue Doppler (p<0.05), and higher TRV at rest (p<0.005).We concluded that patients with SCA and normal PP at rest may exhibit exercise-induced PH, which was related to renal function, increased cardiac chambers, abnormal indices of diastolic function and baseline TRV levels. The clinical meaning of these findings requires clarification in future studies.

ELIGIBILITY:
Inclusion Criteria:

* patients with Sickle Cell Anemia homozygous to hemoglobin S
* preserved physical capacity
* steady state of the disease

Exclusion Criteria:

* Pulmonary Hypertension at rest
* Recent sickling crisis(<2 months)
* High Blood Pressure
* Atrial fibrillation
* Chronic obstructive pulmonary disease
* Last blood transfusion > 3 months before
* Signs of congestive heart failure or significant valve disease
* Normal global and regional systolic function on echocardiography

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with SCA, homozygous to hemoglobin S with preserved physical capacity, followed at the Hematology and Blood Transfusion Division of the Federal University of Sao Paulo (UNIFESP) or at the Hematology and Oncology Division of Santa Casa de Misericordia de Sao Paulo Medical School.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2006-06; Primary Completion 2006-12 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Exercise-induced pulmonary hypertension | until one minute after exercise

CONTACTS AND LOCATIONS:
Overall Officials: Orlando C Filho, Study Chair — Federal University of São Paulo